CLINICAL TRIAL: NCT05263492
Title: A Multicenter, Open-Label Phase 2 Study to Evaluate the Safety and Efficacy of Lenvatinib in Combination With Pembrolizumab in Black Participants With Mismatch Repair-Proficient Recurrent Endometrial Cancer
Brief Title: Study of Lenvatinib w/ Pembro in Black Participants w/Mismatch Repair-Prof Recurrent Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed early due to low enrollment rates
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21-18659; HM20023447 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer; Mismatch Repair-Proficient; Recurrent Endometrial Cancer
Keywords: Endometrial Cancer; Mismatch Repair-Proficient; Recurrent; Lenvatinib; Black Participants; Pembrolizumab
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab & Lenvatinib (Experimental): Lenvatinib, 20 mg administered orally (PO) once daily (QD) during each 21-day cycle, and Pembrolizumab, 200 mg administered by intravenous (IV) infusion on day 1 of each 21-day cycle.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib once a day by mouth every day
Drug: Pembrolizumab — Pembrolizumab through a needle or tube in a vein (intravenously, IV) every 3 weeks.

SUMMARY:
Determine the efficacy of the combination of lenvatinib and pembrolizumab in Black participants

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multicenter phase 2 trial designed to prospectively evaluate the safety and efficacy of lenvatinib in combination with pembrolizumab for mismatch repair proficient recurrent endometrial cancer in Black patients (a population under-represented on 2 FDA registration trials).

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed endometrioid, serous, clear cell, carcinosarcoma, or de-differentiated or undifferentiated endometrial cancer with radiographic and/or clinical evidence of disease progression
* Documented microsatellite stable disease as tested by either microsatellite instability polymerase chain reaction (MSI PCR) or deoxyribonucleic acid (DNA) mismatch repair (MMR) by immunohistochemistry (IHC)
* Self-identify as being of predominantly (>50%) Black race, inclusive of Black, African-American, Black Hispanic (Afro-Latinx), African, or Afro-Caribbean ancestry
* Received, ineligible for (by investigator determination), or declined platinum containing chemotherapy
* Received no greater than two prior lines of therapy. Maintenance therapies and hormonal therapies will NOT count as a line of therapy.
* Measurable disease as determined by RECIST v1.1:
* At least one lesion of ≥10 mm in the longest diameter for a non-lymph node, or ≥15 mm in the short-axis diameter for a lymph node that is serially measurable using computerized tomography/magnetic resonance imaging (CT/MRI)
* Target lesions limited to a radiated field must show evidence of substantial size increase according to previous scans to be deemed a target lesion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Ability to swallow oral medications
* Patients who are not postmenopausal or have not undergone hysterectomy must have a documented negative serum pregnancy test within 72 hours prior to initiating study treatment

Note: Postmenopausal is defined as any of the following:

* Age ≥ 60 years
* Age < 60 years and amenorrheic for at least 1 year with follicle-stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range
* Bilateral oophorectomy
* Patients of child-bearing potential must agree to use a medically accepted method for preventing pregnancy during and for a minimum of 4 months following the last dose of lenvatinib or pembrolizumab
* Patients with known brain metastases will be eligible if they have completed primary brain therapy (such as whole brain radiotherapy, stereotactic radiosurgery, or complete surgical resection) and if they have remained clinically stable, asymptomatic, and off of steroids for at least 28 days before starting study treatment
* Toxicities from previous cancer therapies resolved to grade ≤1 unless specified otherwise (exceptions: chronic residual toxicities that in the opinion of the investigator are not clinically relevant, given the known safety/toxicity profiles of Lenvatinib and pembrolizumab, such as alopecia, grade ≤2 anemia; neuropathy related to previous chemotherapy must be resolved to grade ≤2)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Carcinosarcoma (malignant mixed mullerian tumor), endometrial leiomyosarcoma, or endometrial stromal sarcoma
* Unstable central nervous system (CNS) metastases
* Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib
* Pre-existing grade ≥3 gastrointestinal or non-gastrointestinal fistula
* Radiographic evidence of major blood vessel invasion/infiltration
* Clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study treatment
* History of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, cerebrovascular accident, stroke, or cardiac arrhythmia associated with hemodynamic instability within 12 months of the first dose of study treatment
* Known history or evidence of interstitial lung disease or active, non-infectious pneumonitis
* Administration of or condition requiring administration of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating study treatment Exception: Patients with conditions that can be managed with steroids equivalent to or less than an oral prednisone dose of 10 mg daily are not excluded from the study
* Active autoimmune disease (with the exception of psoriasis) that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents Note: Patients with the conditions or medical history listed below are not excluded from the study.

  * Vitiligo
  * Resolved childhood asthma/atopy
  * Requirement for intermittent use of bronchodilators or local steroid injections or topical steroids
  * Hypothyroidism stable on hormone replacement
  * Sjogren's Syndrome
* Has received >1 prior systemic chemotherapy regimen (other than adjuvant or neoadjuvant) for endometrial cancer; participants may receive up to two regimens of platinum-based chemotherapy in total, as long as one is given in the neoadjuvant or adjuvant treatment setting
* Prior anticancer treatment within 28 days of study start
* Prior treatment with any treatment targeting Vascular endothelial growth factor (VEGF)-directed angiogenesis, any anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has received prior treatment with an agent directed to a stimulatory or co-inhibitory T-cell receptor other than an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, and who has discontinued from that treatment due to a grade 3 or higher immune-related adverse event (irAE)
* Has received prior radiation therapy within 21 days of study start with the exception of palliative radiotherapy to bone lesions, which is allowed if completed 2 weeks of study start; participants must have recovered from all radiation-related toxicities and/or complications prior to randomization
* Participants with urine protein ≥3.5 gram (g)/24 hour
* Left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO)
* Prior immunotherapy (single or dual immune checkpoint inhibition, cellular or vaccine therapy)
* Administration of a live vaccine within 30 days prior to initiating study treatment Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are permitted; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed. Coronavirus Disease 2019 (COVID-19) vaccines are allowed and encouraged
* Administration of any investigational agent within 4 weeks prior to initiating study treatment
* History of solid organ or allogeneic stem cell transplant
* Known intolerance to either of the study drugs (or any of the excipients)
* Known immunodeficiency, eg, human immunodeficiency virus (HIV) Note: HIV testing is not required for eligibility screening
* Known active hepatitis B or C Note: hepatitis B and C testing is not required for eligibility screening
* Serious (ie, grade ≥3) uncontrolled infection
* Pregnancy or breastfeeding
* Diagnosis or treatment for another malignancy within 2 years prior to study registration, with the following exceptions: complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, any in situ malignancy
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea Salyer, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data to other researchers at this time.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab & Lenvatinib
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Disease progression during active treatment | 3

BASELINE CHARACTERISTICS:
Population: The trial was terminated. Only 4 participants were enrolled in this trial. Based on the low enrolment numbers, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Pembrolizumab & Lenvatinib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Determine the Objective Response Rate (ORR) at 24 Weeks in Black Patients With Recurrent Endometrial Cancer Treated With Lenvatinib 20 mg Orally Daily in Combination With Pembrolizumab 200 mg IV Every 3 Weeks
Description: Number of patients evaluable for measurement of tumor response evaluated and recorded according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Time Frame: 24 Weeks
Population: This trial only recruited 4 participants, data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Pembrolizumab & Lenvatinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Determine the Median Progression Free Survival (PFS)
Description: Number of patients who are alive following last dose of study treatment
Time Frame: Up to 90 days following the last dose of study treatment
Population: Only 4 participants were enrolled on this protocol, data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Pembrolizumab & Lenvatinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Determine the Median Progression Free Survival (PFS)
Description: Number of patients who have not had disease progression following last dose of study treatment
Time Frame: Up to 90 days following the last dose of study treatment
Population: The trial was terminated. Only 4 participants were enrolled in this trial, data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Pembrolizumab & Lenvatinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Determine the Median Progression Free Survival (PFS)
Description: Number of patients who have not relapsed following last dose of study treatment
Time Frame: Up to 90 days following the last dose of study treatment
Population: The trial was terminated. Only 4 participants were enrolled, data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Pembrolizumab & Lenvatinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine the Number of Patients With Treatment-related Adverse Events (AEs) in the Study Population
Description: Using criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0), all AEs captured
Time Frame: Up to 30 days following the last dose of study treatment
Population: The trial was terminated. Only 4 participants were enrolled in this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab & Lenvatinib
Number analyzed (Participants) | 4
Participants | 4

6. Secondary Outcome: Determine the Number of Patients Who Discontinue Treatment Due to Treatment-related Adverse Events (AEs)
Description: Number of patients who discontinue treatment due to treatment-related AEs.
Time Frame: up to 30 days (plus or minus 15 days) following last dose of study treatment, average of 4.75 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab & Lenvatinib
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the informed consent form was signed, through end of treatment visit, +/- 15 days after the last administered component of study regimen, and every three months during survival status until patient disease progression, relapse, or death, average of 4.75 months.
Description: The trial was terminated. Only 4 participants were enrolled in this trial.
Arm/Group | Pembrolizumab & Lenvatinib
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab & Lenvatinib (N=4)
Anemia (Blood and lymphatic system disorders) | 3 (9)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (5)
Fatigue (General disorders) | 4 (11)
Fever (General disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (8)
Lymphocyte count decreased (Investigations) | 4 (17)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 3 (3)
Thyroid stimulating hormone increased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Hypertension (Vascular disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
This trial was terminated early for low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT05263492/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT05263492/ICF_000.pdf